CLINICAL TRIAL: NCT00292786
Title: Electrical Stimulation Gait Training to Effect Improvements in Walking Function and Posture for Children With Cerebral Palsy
Brief Title: The Effects of Electrical Stimulation Gait Training on Walking and Posture for Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8520; 4365
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2008-02-05 (Estimated); Status verified 2008-02

CONDITIONS: Cerebral Palsy
Keywords: Functional Electrical Stimulation; FES; Walking; Practice; Coordination; Posture
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Walking Practice with Functional Electrical Stimulation
Behavioral: Walking Practice

SUMMARY:
This proposal is designed to achieve the following specific aims and will test the associated hypotheses:

AIM 1: To compare walking ability, standing posture, gait initiation and functional standing and stepping of twenty children with typical development to that of twenty children with spastic diplegia or hemiplegia, CP.

Hypotheses

* Children with CP will demonstrate impaired coordination as compared to children of typical development. In addition, children with CP will demonstrate inappropriate foot contact area, decreased velocity and step length as compared to children of typical development.
* Children with CP will demonstrate impaired postural control as compared to children of typical development.
* Children with CP will demonstrate an impaired gait initiation motor program as compared to children with typical development.
* Children with CP will take more time to complete the timed up and go test and demonstrate decreased reaching distances in the functional reach test as compared to children of typical development.

AIM 2: Using a single-blinded, randomized, controlled study design, to assess the ability of a 12-week at-home electrical stimulation gait training program to improve walking ability, standing posture, gait initiation, functional standing and stepping, and satisfaction with walking ability for a group of 10 children with spastic diplegia or hemiplegia CP as compared to a group of 10 children with spastic diplegia or hemiplegia CP who undergo a 12-week at-home gait training program without electrical stimulation.

Hypotheses

* The ES gait training group will demonstrate improved joint coordination as compared to the group undergoing a gait training program without ES. The ES gait training group will demonstrate improved foot contact area, increased self-selected walking velocity and greater step length as compared to the group undergoing a gait training program without ES.
* The ES gait training group will demonstrate improved postural control as compared to the group undergoing a gait training program without ES.
* The ES gait training group will demonstrate improved gait initiation as compared to the gait training group without ES.
* The ES gait training group will demonstrate decreased times on the Timed Up and Go and an increase in functional reach as compared to the group undergoing a gait training program without ES.
* The ES gait training group will demonstrate greater satisfaction and self-perceived performance on everyday tasks related to walking function and posture as measured by the COPM compared to the group that undergoes a gait training program without ES.

DETAILED DESCRIPTION:
This is a single blinded, randomized, controlled pre-test/post-test study design (Figure 4). The twenty children with spastic diplegia or hemiplegia CP will be randomized by a statistician to one of two treatment groups. One group will undergo a 12-week at-home gait training program with ES, subjects/guardians can choose either the surface or percutaneous stimulation subgroup, and the second group will undergo a 12-week at-home gait training program without ES. For both groups, data will be collected at five points: just before gait training, after 4 and 8 weeks of gait training, at the conclusion of gait training (after 12 weeks), and 4 weeks after gait training has been discontinued (16 weeks post initiation of gait training). Data collection at each follow-up point will include the kinetics and kinematics of walking, standing posture, gait initiation, plantar pressures, the administration of the Timed Up & Go and Functional Reach Test, and the assessment of lower extremity muscle strength using a hand-held dynamometer. The Canadian Occupational Performance Measure (COPM) will be applied before and after the 12-week gait training program and 4 weeks after the gait training has been discontinued. For the 20 children with typical development, the same data will be collected (except for the COPM) and used for comparison to the pre-training data collected from all 20 children with CP.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of spastic diplegia or spastic hemiplegia or a history of typically development for the measurement only group.
* A Level I, II or III gross motor function classification.
* The subject classified as Level I or II is able to walk indoors and outdoors and climb stairs holding onto a railing but experiences limitations walking in crowds or confined spaces. Subjects classified as Level III's need to walk with assistive devices and have limitations in their ability to ambulate outdoors and in the community. Children have at best only minimal ability to perform gross motor skills such as running and jumping.
* Male or female between the ages of 7 and 14 years of age.
* Family able and willing to provide adequate care to electrodes and electrode sites.
* Must be orthopedically cleared without imminent risk of hip subluxation or dislocation and no significant scoliosis.
* Seizure-free.
* Visuoperceptual skills and cognitive/communication skills sufficient to follow multiple step commands and to attend to tasks associated with data collection.
* Absence of severe tactile hypersensitivity in the lower extremities.
* Willingness to stay in Philadelphia for extended period of time to train and return for follow-up data.
* Written, informed consent.
* One year post soft tissue releases to the lower extremities.
* Passive range of motion of lower extremity joints: <10 degrees contracture of hip in extension as measured by the Thomas Test; <5 degrees knee flexion contracture and popliteal angle <45 degrees; at least 0 degrees of ankle dorsiflexion with knee extended and foot in varus.

Exclusion Criteria:

* Children with "mixed" types of CP (ie:Athetosis) or other movement disorders (ie:Ataxia).
* Allergy or sensitivity to non-latex tape placed in the skin
* Female children cannot be pregnant. A pregnancy test will be given if it is possible that the child can become pregnant, to ascertain whether or not the child is pregnant.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Gait Kinematics, Spatial Temporal Parameters &Interjoint coordination, Standing Center of Pressure Variables, Canadian Occupational Performance Measurement, Muscle activation and timing, Timed up and go test, Functional Reach test

CONTACTS AND LOCATIONS:
Overall Officials: James J McCarthy, MD, Principal Investigator — Shriners Hospital for Children Philadelphia; Carole A Tucker, PhD, PT, Study Director — Shriners Hospital Philadelphia
Locations (1):
- Shriners Hospital for Children Philadelphia, Philadelphia, Pennsylvania, United States